CLINICAL TRIAL: NCT06170021
Title: Effect of Irradiation Dose to Eustachian Tube and Surrounding Auditory Organs on the Occurrence of Radiation-induced Otitis Media in Nasopharyngeal Carcinoma Patients During Intensity Modulated Radiotherapy Era: A Prospective Cohort Study
Brief Title: Occurrence of Radiation-induced Otitis Media in Nasopharyngeal Carcinoma Patients After Intensity Modulated Radiotherapy
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Director of the Department of Nasopharyngeal Carcinoma, Sun Yat-sen University
Other Study IDs: 2023-FXY-228
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; Radiation-induced Otitis Media
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational cohort study to investigate the incidence of radiation-induced otitis media, changes in tubal function and hearing in newly diagnosed nasopharyngeal carcinoma patients without metastasis at multiple time points from baseline to 1 year after radiotherapy.

DETAILED DESCRIPTION:
Patients with newly diagnosed non-metastatic nasopharyngeal carcinoma (AJCC 8th) will be recruited. The incidence of radiation-induced otitis media, eustachian tube function and hearing level in nasopharyngeal carcinoma patients will be prospectively evaluated by magnetic resonance imaging, otoscope, pure tone audiometry, acoustic immittance test and the Eustachian Tube Dysfunction Questionnaire (ETDQ-7) before treatment and serially up to 1 year after radiotherapy. The quality of life of patients will be evaluated before treatment and serially up to 1 year after radiotherapy. The incidence of radiation-induced otitis media, the changes of eustachian tube function and hearing level, together with the influencing factors, in nasopharyngeal carcinoma patients after induction chemotherapy and concurrent chemoradiotherapy will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70, regardless of sex.
* ECOG (Eastern Cooperative Oncology Group) score: 0-1.
* Patients must sign informed consent and be willing, and well understood the objective and procedure of this study.
* Patients with newly histologically confirmed non-keratinizing nasopharyngeal carcinoma, type of WHO II or III, clinical stage I-IVa (according to the 8th American Joint Committee on Cancer [AJCC] edition.
* No radiotherapy or chemotherapy was administered before enrollment.
* Expected survival time ≥ 6 months.

Exclusion Criteria:

* Women in pregnancy or lactation.
* Patients with significantly lower heart, liver, lung, kidney, bone marrow function and other severe medical condition.
* Prior to radiotherapy, there is a clear underlying disease of the eustachian tube or other ear diseases.
* Patients with otitis media before radiotherapy and have no improvement at the end of radiotherapy.
* Patients with history of middle ear, nasal or nasopharyngeal surgery on the affected side.
* Patients combined with congenital cleft palate and other craniofacial abnormalities.
* Patients with histologically confirmed keratinizing nasopharyngeal carcinoma, type of WHO I.
* Patients with recurrence and distant metastasis.
* Patients with radiotherapy or chemotherapy before.
* Age < 18 or age > 70.
* Patients who changed their initial treatment regimen during the observation period due to disease progression (including tumor residual after radiotherapy, tumor recurrence, and new distant metastases).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed non-metastatic nasopharyngeal carcinoma patients.
Sampling Method: Non-Probability Sample
Enrollment: 215 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2025-12-06 (Estimated); Study Completion 2025-12-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of radiation-induced otitis media | 1 year
  Incidence of radiation-induced otitis media will be assessed prospectively before treatment and serially up to 1 year after radiotherapy by magnetic resonance imaging, otoscope, acoustic immittance test and pure tone audiometry.

SECONDARY OUTCOMES:
Effect of the irradiation dose of eustachian tube, tympanum, cochlea, internal auditory tract and vestibule on the occurrence of radiation-induced otitis media | 1 year
  The occurrence of radiation-induced otitis media will be assessed prospectively before treatment and serially up to 1 year after radiotherapy by magnetic resonance imaging, otoscope, acoustic immittance test and pure tone audiometry.
Effect of irradiation dose in the area around of eustachian tube on the severity of ototoxicity after radiotherapy | 1 year
  Severity of ototoxictiy will be assessed prospectively before treatment and serially up to 1 year after radiotherapy by magnetic resonance imaging, otoscope, acoustic immittance test, pure tone audiometry and the Eustachian Tube Dysfunction Questionnaire (ETDQ-7).
Effect of irradiation dose of eustachian tube on hearing injury | 1 year
  The injury of hearing will be assessed prospectively before treatment and serially up to 1 year after radiotherapy by acoustic immittance test and pure tone audiometry.
Effect of different chemoradiotherapy treatment regimens on the occurrence of radiation-induced otitis media | 1 year
  The occurrence of radiation-induced otitis media will be assessed prospectively before treatment and serially up to 1 year after radiotherapy by magnetic resonance imaging, otoscope, acoustic immittance test and pure tone audiometry.
Correlation between radiation-induced otitis media and life quality after radiotherapy | 1 year
  The life quality will be assessed prospectively before treatment and serially up to 1 year after radiotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nasopharyngeal Carcinoma, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen YP, Chan ATC, Le QT, Blanchard P, Sun Y, Ma J. Nasopharyngeal carcinoma. Lancet. 2019 Jul 6;394(10192):64-80. doi: 10.1016/S0140-6736(19)30956-0. Epub 2019 Jun 6. PMID 31178151
- [Background] Emami B, Lyman J, Brown A, Coia L, Goitein M, Munzenrider JE, Shank B, Solin LJ, Wesson M. Tolerance of normal tissue to therapeutic irradiation. Int J Radiat Oncol Biol Phys. 1991 May 15;21(1):109-22. doi: 10.1016/0360-3016(91)90171-y. PMID 2032882
- [Background] Hsin CH, Tseng HC, Lin HP, Chen TH. Post-irradiation otitis media, rhinosinusitis, and their interrelationship in nasopharyngeal carcinoma patients treated by IMRT. Eur Arch Otorhinolaryngol. 2016 Feb;273(2):471-7. doi: 10.1007/s00405-015-3518-8. Epub 2015 Jan 30. PMID 25634060
- [Background] Hsin CH, Chen TH, Liang KL, Tseng HC, Liu WS. Postirradiation otitis media with effusion in nasopharyngeal carcinoma patients treated by intensity-modulated radiotherapy. Laryngoscope. 2013 Sep;123(9):2148-53. doi: 10.1002/lary.23215. Epub 2013 Jul 8. PMID 23835775
- [Background] Yao JJ, Zhou GQ, Lin L, Zhang WJ, Peng YL, Chen L, Tang LL, Mao YP, Ma J, Sun Y. Dose-volume factors associated with ear disorders following intensity modulated radiotherapy in nasopharyngeal carcinoma. Sci Rep. 2015 Sep 1;5:13525. doi: 10.1038/srep13525. PMID 26323586
- [Background] Wang SZ, Wang WF, Zhang HY, Guo M, Hoffman MR, Jiang JJ. Analysis of anatomical factors controlling the morbidity of radiation-induced otitis media with effusion. Radiother Oncol. 2007 Dec;85(3):463-8. doi: 10.1016/j.radonc.2007.10.007. Epub 2007 Nov 19. PMID 18006095